CLINICAL TRIAL: NCT00002691
Title: LSA5 PROTOCOL FOR THE TREATMENT OF ADVANCED PEDIATRIC AND ADOLESCENT NON-HODGKIN'S LYMPHOMA (NHL)
Brief Title: Combination Chemotherapy in Treating Pediatric Patients With Stage III or IV Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 95-065; CDR0000064426 (Registry Identifier: PDQ (Physician Data Query)); NCI-V95-0763
Record Dates: First submitted 1999-11-01; First posted 2004-07-01 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma
Keywords: stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; stage III childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma
MeSH Terms: conditions — Lymphoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating | interventions — Filgrastim; Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Etoposide; Leucovorin; Mesna; Methotrexate; Vincristine

INTERVENTIONS:
Biological: filgrastim
Drug: asparaginase
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: etoposide
Drug: leucovorin calcium
Drug: mesna
Drug: methotrexate
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and using drugs in different ways may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating pediatric patients with stage III or stage IV non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the feasibility of treating all histologic subgroups of pediatric non-Hodgkin's lymphoma on one protocol, with the addition of asparaginase during the induction and consolidation phases for diffuse lymphoblastic lymphoma and T-cell, large noncleaved cell diffuse lymphoma. II. Assess whether intensification of cyclophosphamide during induction therapy will achieve a complete response rate of 95% in 1 to 1.5 months for all histologies. III. Assess whether achieving remission induction in 1 month, administering cytarabine/methotrexate by continuous infusion during consolidation therapy, and increasing the number of intrathecal methotrexate injections throughout protocol therapy decreases central nervous system relapse in these patients. IV. Assess whether a 5-year recurrence-free survival of 85% is achievable for all histologies on this protocol. V. Assess whether duration of maintenance chemotherapy may be stratified by stage and histology of disease to avoid unnecessarily prolonged chemotherapy.

OUTLINE: The following acronyms are used: ARA-C Cytarabine, NSC-63878 ASP Asparaginase, NSC-109229 CF Leucovorin, NSC-3590 CTX Cyclophosphamide, NSC-26271 DM Dexamethasone, NSC-34521 DNR Daunorubicin, NSC-82151 G-CSF Granulocyte Colony-Stimulating Factor, NSC-614629 LBL Lymphoblastic Lymphoma LCALKi1B Large Cell Anaplastic B-cell Lymphoma LCALKi1T Large Cell Anaplastic T-cell Lymphoma LCL Large Cell Lymphoma Mesna Mercaptoethane Sulfonate, NSC-113891 MTX Methotrexate, NSC-740 TMP-SMX Trimethoprim-Sulfamethoxazole VCR Vincristine, NSC-67574 VP-16 Etoposide, NSC-141540 Induction: 2-Drug Combination Systemic Chemotherapy plus Single-Agent Intrathecal Chemotherapy followed by 2- or 3-Drug Combination Systemic Chemotherapy plus Single-Agent Intrathecal Chemotherapy. Part I: CTX/DNR; plus IT ARA-C; followed by Part II: DM/VCR; plus ASP for patients with LBL, T-cell LCL, or LCALKi1T; plus IT MTX. Consolidation: 2- or 3-Drug Combination Systemic Chemotherapy with Leucovorin Rescue followed by 2- or 3-Drug Combination Systemic Chemotherapy. Part I: ARA-C/MTX with CF; plus ASP for patients with LBL, T-cell LCL, or LCALKi1T; followed by Part II: ARA-C/VP-16; plus, for patients with LBL, T-cell LCL, or LCALKi1T. Maintenance. Single-Agent Systemic Chemotherapy with Leucovorin Rescue plus Single-Agent Intrathecal Chemotherapy followed sequentially by 3 2-Drug Combination Systemic Chemotherapy Regimens. Part I: MTX; with CF; plus IT MTX; followed by Part II: CTX/VCR; followed by Part III: ARA-C/VP-16; followed by Part IV: DNR/DM.

PROJECTED ACCRUAL: 25 patients/stratum are expected to be accrued over 3 years. This study will be reviewed for early closure if more than 1 patient has PD.

ELIGIBILITY:
DISEASE CHARACTERISTICS: See General Eligibility Criteria

PATIENT CHARACTERISTICS: See General Eligibility Criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1995-08; Primary Completion 2000-06 (Actual); Study Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Trippett, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States